CLINICAL TRIAL: NCT02619812
Title: A Randomized, Placebo-Controlled, Pilot Study of Colesevelam and Serum-Derived Bovine Immunoglobulin/Protein Isolate to Manage Diarrhea in Patients With Multiple Myeloma Receiving Conditioning Chemotherapy for Autologous Stem Cell Transplantation (SCT)
Brief Title: Manage Diarrhea in Patients With Multiple Myeloma While Receiving Conditioning Chemotherapy for Autologous SCT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty recruiting; pill burden and nausea were barriers
Sponsor: Mayo Clinic (Other)
Collaborators: Entera Health, Inc (Industry)
Responsible Party: Principal Investigator, Michael Camilleri, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 15-006205
Record Dates: First submitted 2015-11-19; First posted 2015-12-02 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Colesevelam Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group A: SBI + Placebo (Active Comparator): Serum-derived bovine immunoglobulin/protein isolate (SBI) 10 grams + placebo twice per day
  Interventions: Other: Serum-derived bovine immunoglobulin/protein isolate (SBI); Other: Double Placebo
- Group B: Colesevelam + Placebo (Active Comparator): Colesevelam 1.875 g + Placebo twice per day
  Interventions: Drug: Colesevelam; Other: Double Placebo
- Group C: Colesevelam + SBI (Active Comparator): Colesevelam 1.875 g + Serum-derived bovine immunoglobulin/protein isolate (SBI) 10 grams twice per day
  Interventions: Other: Serum-derived bovine immunoglobulin/protein isolate (SBI); Drug: Colesevelam
- Group D: Double Placebo (Placebo Comparator): Double placebo twice per day
  Interventions: Other: Double Placebo

INTERVENTIONS:
Other: Serum-derived bovine immunoglobulin/protein isolate (SBI) — SBI 10 grams (The subject will take a total of 4 packets of SBI; taken as two packets of SBI twice a day mixed with water or blended with certain foods)
  Arms: Group A: SBI + Placebo; Group C: Colesevelam + SBI
Drug: Colesevelam — Colesevelam 1.875 g (The subject will take a total of 12 capsules of Welchol 1.875g per day; taken as 6 capsules twice a day by mouth).
  Other Names: Welchol
  Arms: Group B: Colesevelam + Placebo; Group C: Colesevelam + SBI
Other: Double Placebo — Double placebo twice per day (The subject will take a total of 4 packets of placebo and 12 capsules daily taken as 6 capsules twice a day by mouth and two packets of placebo twice a day mixed with water or blended with certain foods).
  Arms: Group A: SBI + Placebo; Group B: Colesevelam + Placebo; Group D: Double Placebo

SUMMARY:
For patients who receive a hematopoietic cell transplant (HCT), there is a risk of developing a diarrhea secondary to the chemotherapy which we give. Diarrhea is usually harmless in healthy adults; however, in transplant patients, diarrhea can result in dehydration, negative impact on quality of life, and prolonged hospitalization. The purpose of this study was to see if Colesevelam (Welchol) and Serum-derived bovine immunoglobulin-protein (SBI) result in a change in the frequency or consistency of your bowel movements.

DETAILED DESCRIPTION:
This was a randomized, double-blind, placebo-controlled pilot study of SBI, colesevelam, and placebo in patients undergoing autologous HSCT for the clinical care of multiple myeloma.

The number of adults undergoing hematopoietic stem cell transplant (HSCT) has grown significantly over the past two decades as a result of the availability of therapies for advanced hematologic and solid tumor malignancies, and the broader selection criteria for eligibility to receive these transplants. Generally, the stem cell transplant procedure consists of administration of chemotherapy and/or radiation therapy to ablate all residual malignancy (called conditioning therapy), followed by intravenous infusion of hematopoietic stem cells to restore bone marrow function. Generally, HSCT has a positive effect on survival, despite serious adverse effects and life-threatening complications.

Diarrhea can affect up to 91% of patients receiving autologous or allogeneic HSCT and is identified by 9% of the patients as the single most debilitating adverse effect post-HSCT. Other commonly encountered symptoms are nausea and vomiting (13%) and mouth sores (42%). The impact of diarrhea can be significant and result in dehydration, negative impact on quality of life, prolonged hospitalization with an increased cost and risk, and the diarrhea may be potentially life-threatening.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, male or female
* Diagnosis: multiple myeloma undergoing Autologous Stem Cell Transplantation (SCT)
* Planning to receive conditioning chemotherapy (Melphalan) for autologous stem cell transplantation and standard prophylactic antibiotics treatment.
* Can drink 200ml of mannitol and agrees to undergo stool, urine, and blood checks 3 times during the study.
* Agrees and able to take the investigational products or placebo starting from the day of completing conditioning therapy for a total of 4 weeks

Exclusion Criteria:

* Patients with history of inflammatory bowel disease will be excluded from the study.
* Patients with prior GI tract surgical (small or large bowel) resections
* The concurrent presence of systemic light chain amyloidosis
* Subject has known allergy or intolerance to beef or to any ingredient used in the product
* Women who are pregnant, breast-feeding and of child-bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subjects were recruited from Mayo Clinic in Rochester, Minnesota.
Pre-assignment Details: A total of 4 subjects were enrolled. Two subjects were randomized to placebo/placebo, and one subject was randomized to colesevelam/Serum-derived bovine immunoglobulin/protein isolate (SBI). One subject was consented, but never randomized/accrued.
Groups:
- Group A: SBI + Placebo: SBI 10 grams + placebo twice per day.
- Group C: Colesevelam + SBI: Colesevelam 1.875 g + SBI 10 grams twice per day.
- Group D: Double Placebo: Double Placebo: Double placebo twice per day (Subjects took a total of 4 packets of placebo and 12 capsules daily taken as 6 capsules twice a day by mouth and two packets of placebo twice a day mixed with water or blended with certain foods).
Period: Overall Study
Arm/Group | Group A: SBI + Placebo | Group B: Colesevelam + Placebo | Group C: Colesevelam + SBI | Group D: Double Placebo
Started | 0 | 0 | 1 | 2
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: SBI + Placebo | Group B: Colesevelam + Placebo | Group C: Colesevelam + SBI | Group D: Double Placebo | Total
Number analyzed (Participants) | 0 | 0 | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  |  | 0 | 0 | 0
  Between 18 and 65 years |  |  | 1 | 2 | 3
  >=65 years |  |  | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  |  | 0 | 0 | 0
  Male |  |  | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States |  |  | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Stool Frequency
Description: Stool frequency was self reported in a daily bowel pattern diary for 30 days.
Time Frame: 30 days
Population: Data were not collected.
Arm/Group | Group A: SBI + Placebo | Group B: Colesevelam + Placebo | Group C: Colesevelam + SBI | Group D: Double Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Primary Outcome: Stool Consistency
Description: The subjects rated their stool consistency using the Bristol Stool Scale. The Bristol Stool Scale is a medical aid designed to classify the form of human feces into seven categories or types. Types 1 and 2 indicate constipation with 3 and 4 being the "ideal stools" especially the latter, as they are the easiest to defecate, and 5-7 tending towards diarrhea.
Time Frame: 30 days
Population: Data were not collected.
Arm/Group | Group A: SBI + Placebo | Group B: Colesevelam + Placebo | Group C: Colesevelam + SBI | Group D: Double Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Group A: SBI + Placebo | Group B: Colesevelam + Placebo | Group C: Colesevelam + SBI | Group D: Double Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 1/1 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: SBI + Placebo (N=0) | Group B: Colesevelam + Placebo (N=0) | Group C: Colesevelam + SBI (N=1) | Group D: Double Placebo (N=2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomach cramps (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was terminated early due to difficulty recruiting subjects; pill burden and nausea were barriers to study continuation for subjects accrued. Data were not collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes